CLINICAL TRIAL: NCT06460922
Title: 3D Printing Models and Personalized Guides in Surgical Planning of Shortening, Wedge and Dorsolateral Biplane Closing Osteotomies in Kienbock´s Disease Stages II and III.
Brief Title: 3D Printing Models in Surgical Planning of Osteotomies in Kienbock´s Disease Stages II-III
Status: Recruiting | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-MPG-2024-04
Record Dates: First submitted 2024-05-21; First posted 2024-06-14 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-03

CONDITIONS: Kienbock Disease
Keywords: Lunatomalacia; Kienböck´s disease; Radial osteotomy; Biplane radial osteotomy
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Radial osteotomy — 3D printing models and personalized guides in surgical planning in distal radius osteotomies for Kienböck´s disease. Osteosynthesis with a plate in distal radius.

SUMMARY:
Ischemic necrosis of lunate bone, osteonecrosis or Kienböck´s disease was described by Kienböck in 1910. Numerous surgical procedures for this disease had been proposed. These surgical options, that depends of the radiological stage and anatomical risk factors, can be classified into lunate unloading procedures, lunate revascularization, replacement procedures and salvage procedures. These procedures, except the salvage procedures, has been successful in reconstructing and maintaining the height of the carpus, avoiding progression of the disease and with reduction of the pain.

The lunate unloading procedures are surgical treatments that make a radial osteotomy for modify differents anatomical risk factors associated with the osteonecrosis.

DETAILED DESCRIPTION:
The anatomical factors associated with Kienböck´s disease are morphology of the lunate type I by Antuña-Zapico, cubitus minus, radial inclination angle greater than 23º, and little coverage of the lunate by the radius.

The types of radial osteotomy for Kienböck´s disease stages II, IIIA, IIIB or IIIC, depends to the anatomy of the patient and its anatomical risk factors. For patients with cubitus minus the indication is usually a radial shortening osteotomy. For patients with zero variant and an increase in the radial inclination angle the indication is usually a closed wedge radial osteotomy. The dorsolateral biplane radial osteotomy is used for zero variant cases such as a modification of the technique proposed by Nakamura et and Miura et al. It decompresses the lunate on the frontal plane and reduces dorsal radiolunate impingement on hyperextension. Dorsolateral radial osteotomy ensures a reduction of the radial inclination angle and a corresponding lunate decompression on the anteroposterior and sagittal plane.

ELIGIBILITY:
Inclusion Criteria:

* Kienbock´s disease in the wrist estages II, IIIA, IIIB or IIIC by Lichtman classification

Exclusion Criteria:

* Pre-radiological stages-Lichtman stage I
* Radiocarpal and midcarpal osteoarthrosis, Lichtman stage IV
* Kienböck in children: less than 18 years
* Adults years greater than 85 years old

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients affected by lunate necrosis of the wrist, lunatomalacia, or Kienböck´s disease, stages II, IIIA, IIIB or IIIC by Lichtman classification, in which a distal radial osteotomy is indicated.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation preoperative and postoperative: Mayo Wrist Score | 22 months
  Modified Mayo Wrist Score (MWS). It is based on pain, range of motion, grip strength and function. Scores of 80 to 100 are considered excellent; 65 to 79, good; 50 to 64, moderate; and less than 50, poor.
Disabilities of the arm, shoulder and hand score questionnaire | 22 months
  Disabilities of the arm, shoulder and hand score (Quick DASH) questionnaire. From 0 (better outcome) to 100% (worse outcome)
Clinical evaluation preoperative and postoperative: Grip strength | 22 months
  Grip strength mesure with a Jamar dynamometer (in Kilograms).
Radiological variables In the posteroanterior radiographs wrist: Lichtman classification | 22 months
  Lichtman´s Stage of lunate necrosis classification: 4 stages (1977). Better stage 1, worse stage 4.
Radiological variables In the posteroanterior radiographs wrist: Carpal Ulnar Distance Ratio. | 22 months
  Carpal Ulnar Distance Ratio (mesure in millimeters) by McMurtry-Youm (1978). Outcomes in a ratio 0.30+-0.03.
Radiological variables In the posteroanterior radiographs wrist. Carpal Height Ratio. | 22 months
  Carpal Height Ratio (measure in millimeters) by McMurtry-Youm (1978) . Outcomes in a ratio 0.54+-0.03.
Radiological variables In the posteroanterior radiographs wrist: Radial Inclination Angle. | 22 months
  The Radial Inclination Angle (RIA) describes the angulation of the distal radial articular surface in relationship with the long axis of the radius or ulna as seen in the posteroanterior view of the wrist. We measure RIA in relationship with the long axis of the ulna. The normal limits are 18.8° to 29.3° (measure in degrees).
Radiological variables In the posteroanterior radiographs wrist: Lunate covering Ratio. | 22 months
  The Lunate Covering Ratio (LCR) is a measure of the lunate surface protected by the radius, obtained by dividing the width of lunate covered by radius by total lunate width in millimeters x 100.
Radiological variables In the posteroanterior radiographs wrist. Ulnar Variance. | 22 months
  Ulnar variance was measured as described by Gelberman et al. (1980) The measurement was obtained by projecting a line from the carpal joint surface of the distal end of the radius toward the ulna and measuring the distance in millimeters between this line and the carpal surface of the ulna. Ulnar shortening values of 2 or more millimeters are described as negative ulna or cubitus minus. Zero variant or neutral ulna with ulnar variance or distal radio-ulnar index is between 0-2 mm and cubitus plus when ulnar elongation values greater than 2 mm.
Clinical evaluation preoperative and postoperative: Pain | 22 months
  Visual Analog Score, from 0 to 10. Better outcome 0 and worse 10.
Clinical evaluation preoperative and postoperative: Range of motion | 22 months
  Range of motion (ROM): wrist motion (flexion, extension, radial deviation, ulnar deviation, pronation, supination) mesure with a goniometer (in degrees).

SECONDARY OUTCOMES:
Radiological variables in the lateral radiograph in the wrist: Palmar Tilt | 22 months
  Palmar tilt (PT) measure in degrees. Palmar tilt is determined by the line drawn across the most distal points of the dorsal and ventral rims of the distal articular surface. The degree of PT is derived by the intersection of the line of PT and a line perpendicular to the long axis of the radius, as seen in the lateral view. The normal limits are 0° to 18°.
Radiological variables in the lateral radiograph in the wrist: Stahl´s Index | 22 months
  Stahl´s index measures the degree of lunate fragmentation and collapse. The normal limits are 0.53+- 0.03. The longitudinal height of the lunate measured on the lateral view is divided by its greatest dorsopalmar dimension. The ratio of these 2 measurements gives the Stahl index.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Lamas, MD, Ph D, Principal Investigator — Research Institute IIB Sant Pau. Institut de Recerca de l´Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
No plan to share

REFERENCES:
- [Result] Calfee RP, Van Steyn MO, Gyuricza C, Adams A, Weiland AJ, Gelberman RH. Joint leveling for advanced Kienbock's disease. J Hand Surg Am. 2010 Dec;35(12):1947-54. doi: 10.1016/j.jhsa.2010.08.017. Epub 2010 Oct 25. PMID 20971577
- [Result] Horii E, Garcia-Elias M, Bishop AT, Cooney WP, Linscheid RL, Chao EY. Effect on force transmission across the carpus in procedures used to treat Kienbock's disease. J Hand Surg Am. 1990 May;15(3):393-400. doi: 10.1016/0363-5023(90)90049-w. PMID 2348055
- [Result] Kennedy C, Abrams R. In Brief: The Lichtman Classification for Kienbock Disease. Clin Orthop Relat Res. 2019 Jun;477(6):1516-1520. doi: 10.1097/CORR.0000000000000595. No abstract available. PMID 30507834
- [Result] Lamas C, Mir X, Llusa M, Navarro A. Dorsolateral biplane closing radial osteotomy in zero variant cases of Kienbock's disease. J Hand Surg Am. 2000 Jul;25(4):700-9. doi: 10.1053/jhsu.2000.6929. PMID 10913211
- [Result] Lamas C, Carrera A, Proubasta I, Llusa M, Majo J, Mir X. The anatomy and vascularity of the lunate: considerations applied to Kienbock's disease. Chir Main. 2007 Feb;26(1):13-20. doi: 10.1016/j.main.2007.01.001. Epub 2007 Feb 8. PMID 17418764
- [Result] Nakamura R, Watanabe K, Tsunoda K, Miura T. Radial osteotomy for Kienbock's disease evaluated by magnetic resonance imaging. 24 cases followed for 1-3 years. Acta Orthop Scand. 1993 Apr;64(2):207-11. doi: 10.3109/17453679308994572. PMID 8498188
- [Result] Matsushita K, Firrell JC, Tsai TM. X-ray evaluation of radial shortening for Kienbock's disease. J Hand Surg Am. 1992 May;17(3):450-5. doi: 10.1016/0363-5023(92)90346-q. PMID 1613218
- [Result] Miura H, Sugioka Y. Radial closing wedge osteotomy for Kienbock's disease. J Hand Surg Am. 1996 Nov;21(6):1029-34. doi: 10.1016/s0363-5023(96)80311-x. PMID 8969427
- [Result] Trumble T, Glisson RR, Seaber AV, Urbaniak JR. A biomechanical comparison of the methods for treating Kienbock's disease. J Hand Surg Am. 1986 Jan;11(1):88-93. doi: 10.1016/s0363-5023(86)80111-3. PMID 3944452
- [Result] Tsuge S, Nakamura R. Anatomical risk factors for Kienbock's disease. J Hand Surg Br. 1993 Feb;18(1):70-5. doi: 10.1016/0266-7681(93)90201-p. PMID 8436868
- [Result] Soejima O, Iida H, Komine S, Kikuta T, Naito M. Lateral closing wedge osteotomy of the distal radius for advanced stages of Kienbock's disease. J Hand Surg Am. 2002 Jan;27(1):31-6. doi: 10.1053/jhsu.2002.30906. PMID 11810611
- [Result] Watanabe K, Nakamura R, Horii E, Miura T. Biomechanical analysis of radial wedge osteotomy for the treatment of Kienbock's disease. J Hand Surg Am. 1993 Jul;18(4):686-90. doi: 10.1016/0363-5023(93)90319-X. PMID 8349982
- [Result] Werner FW, Palmer AK. Biomechanical evaluation of operative procedures to treat Kienbock's disease. Hand Clin. 1993 Aug;9(3):431-43. PMID 8408253
- [Result] Ma ZJ, Liu ZF, Shi QS, Li T, Liu ZY, Yang ZZ, Liu YH, Xu YJ, Dai K, Yu C, Gan YK, Wang JW. Varisized 3D-Printed Lunate for Kienbock's Disease in Different Stages: Preliminary Results. Orthop Surg. 2020 Jun;12(3):792-801. doi: 10.1111/os.12681. Epub 2020 May 17. PMID 32419366